CLINICAL TRIAL: NCT06915298
Title: Impact of Providing Health Information on Alcohol Labels in a Real-World Setting: a Randomized Controlled Trial Among Supermarket Customers in Barcelona
Brief Title: Impact of Alcohol Labels in a Real-World Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: World Health Organization (Other)
Collaborators: IPSOS (Industry); Program on Substance Abuse, Public Health Agency, Government of Catalonia (Unknown)
Responsible Party: Principal Investigator, Daša Kokole, Principal Investigator, World Health Organization
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ERC.0004213; 24/228-P (Other: Ethical Committee for Research with Medicines (CEIm) IDIAP Jordi Gol)
Record Dates: First submitted 2025-04-01; First posted 2025-04-08 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Knowledge; Behaviour Change; Risk Perception; Intention; Support for Alcohol Policies; Emotional Response; Product Appeal
Keywords: alcohol; health warning label; supermarket
MeSH Terms: interventions — Ethanol; Drug Labeling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Responsibility message - front of the container / no pre-test (Active Comparator): A sticker with a message to drink responsibly is applied to the front of the container.
  There is no question on knowledge of alcohol related harms at baseline.
  Interventions: Behavioral: Responsibility message on alcohol label; Behavioral: Front label; Other: No outcome pre-testing
- Responsibility message - back of the container / no pre-test (Active Comparator): A sticker with a message to drink responsibly is applied to the back of the container.
  There is no question on knowledge of alcohol related harms at baseline.
  Interventions: Behavioral: Responsibility message on alcohol label; Behavioral: Back label; Other: No outcome pre-testing
- Cancer message - front of the container / no pre-test (Experimental): A sticker with a message on alcohol causing cancer is applied to the front of the container.
  There is no question on knowledge of alcohol related harms at baseline.
  Interventions: Behavioral: Alcohol health warning label - cancer; Behavioral: Front label; Other: No outcome pre-testing
- Cancer message - back of the container / no pre-test (Experimental): A sticker with a message on alcohol causing cancer is applied to the back of the container.
  There is no question on knowledge of alcohol related harms at baseline.
  Interventions: Behavioral: Alcohol health warning label - cancer; Behavioral: Back label; Other: No outcome pre-testing
- Responsibility message - front of the container / pre-test (Active Comparator): A sticker with a message to drink responsibly is applied to the front of the container. There is a question on knowledge of alcohol related harms at baseline.
  Interventions: Behavioral: Responsibility message on alcohol label; Behavioral: Front label; Other: Outcome pre-testing
- Responsibility message - back of the container / pre-test (Active Comparator): A sticker with a message to drink responsibly is applied to the back of the container. There is a question on knowledge of alcohol related harms at baseline.
  Interventions: Behavioral: Responsibility message on alcohol label; Behavioral: Back label; Other: Outcome pre-testing
- Cancer message - front of the container / pre-test (Experimental): A sticker with a message on alcohol causing cancer is applied to the front of the container. There is a question on knowledge of alcohol related harms at baseline.
  Interventions: Behavioral: Alcohol health warning label - cancer; Behavioral: Front label; Other: Outcome pre-testing
- Cancer message - back of the container / pre-test (Experimental): A sticker with a message on alcohol causing cancer is applied to the back of the container. There is a question on knowledge of alcohol related harms at baseline.
  Interventions: Behavioral: Alcohol health warning label - cancer; Behavioral: Back label; Other: Outcome pre-testing

INTERVENTIONS:
Behavioral: Alcohol health warning label - cancer — A sticker with health information on alcohol causing cancer is applied to alcoholic beverage containers purchased by the participants.
  Arms: Cancer message - back of the container / no pre-test; Cancer message - back of the container / pre-test; Cancer message - front of the container / no pre-test; Cancer message - front of the container / pre-test
Behavioral: Responsibility message on alcohol label — A sticker with a message to drink responsibly will be applied to alcoholic beverage containers purchased by the participants.
  Arms: Responsibility message - back of the container / no pre-test; Responsibility message - back of the container / pre-test; Responsibility message - front of the container / no pre-test; Responsibility message - front of the container / pre-test
Behavioral: Front label — A sticker will be applied to the front of the alcoholic beverage containers purchased by the participants.
  Arms: Cancer message - front of the container / no pre-test; Cancer message - front of the container / pre-test; Responsibility message - front of the container / no pre-test; Responsibility message - front of the container / pre-test
Behavioral: Back label — A sticker will be applied to the back of the alcoholic beverage containers purchased by the participants.
  Arms: Cancer message - back of the container / no pre-test; Cancer message - back of the container / pre-test; Responsibility message - back of the container / no pre-test; Responsibility message - back of the container / pre-test
Other: Outcome pre-testing — Primary outcome (knowledge of alcohol related harms) is tested at baseline.
  Arms: Cancer message - back of the container / pre-test; Cancer message - front of the container / pre-test; Responsibility message - back of the container / pre-test; Responsibility message - front of the container / pre-test
Other: No outcome pre-testing — Primary outcome (knowledge of alcohol related harms) is not tested at baseline.
  Arms: Cancer message - back of the container / no pre-test; Cancer message - front of the container / no pre-test; Responsibility message - back of the container / no pre-test; Responsibility message - front of the container / no pre-test

SUMMARY:
The goal of this randomized controlled trial is to evaluate the impact of health information labeling on alcohol-related knowledge and behaviors in adults purchasing alcohol in Barcelona, Spain. The main questions it aims to answer are:

* Does a label containing a cancer message have a larger impact on knowledge, behavior, intentions, risk perception, emotional response, product appeal and policy support compared to a responsibility label?
* Does the positioning of the label (front vs. back) on the alcohol container affect these outcomes?

Researchers will compare the impact of cancer message labels vs. responsibility labels and front vs. back positioning to see if there are differences in the primary outcome (knowledge of alcohol causing cancer) and secondary outcomes (behavior, intentions, risk perception, emotional response, and policy support).

Additionally, the study will provide insight in whether there is a testing effect of primary outcome pre-measurement by exposing only half of the sample to baseline question on knowledge of alcohol related harms.

Participants will:

* Be recruited in front of selected supermarkets in Barcelona after purchasing alcohol for their own consumption.
* Complete a baseline questionnaire.
* Receive a sticker containing a randomly assigned health message that will be applied to every alcohol beverage they have purchased.
* Receive an invitation to complete two follow-up surveys, one a week and one a month after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* have just purchased at least one alcoholic beverage container for their own consumption
* speak Spanish or Catalan
* are 18 years or older
* provide informed consent to participation

Exclusion Criteria:

- all the purchased alcohol containers are too small for a label sticker to be affixed

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1410 (Actual)
Dates: Start 2025-04-23 (Actual); Primary Completion 2025-07-25 (Actual); Study Completion 2025-07-25 (Actual)

PRIMARY OUTCOMES:
Knowledge of alcohol causing cancer | 1 week / 1 month
  Knowledge will be assessed with the question "Which of the following diseases and conditions does alcohol consumption increase the risk of? (select all that apply)", with the possible choices being "Cancer", "Heart disease", "Respiratory disease", "Alcohol Use Disorder", "Injuries", "Diabetes" and "Liver disease" displayed randomly, and "I don't know" and "None" as exclusive options. If participants select "Cancer" as an outcome, a follow up question will ask: "Which of the following cancers do you think drinking alcohol increases the risk of? (select all that apply)", with "Female breast cancer", "Liver cancer", "Colon cancer", "Skin cancer", "Oral cancer", displayed randomly, and "I don't know" and "None" as exclusive options. The outcome will be dichotomous based on whether the participants correctly identify the link between alcohol and two cancers mentioned in the label: breast and colon cancer.

SECONDARY OUTCOMES:
Alcohol consumption behaviour | 1 week / 1 month
  Decrease in alcohol consumption will be measured with measuring the amount of standard drinks consumed in the last 7 days ("How many standard drinks of alcohol did you drink over the last 7 days?"), as well as based on question on whether they have foregone an alcoholic drink because they wanted to drink less (In the last 7 days, did you ever forego an alcoholic drink because you wanted to drink less? Yes/No).
Risk perception | 1 week / 1 month
  Perceived personal cancer risk will be measured with question "If I consume alcohol on a regular basis, I am at greater risk of getting cancer." Perceived general health risk will be measured with question "If I consume more alcohol, I am at greater risk for health harm". Both questions will be measured on 5-point Likert scale (strongly Disagree to Strongly Agree).
Behavioural intention | 1 week / 1 month
  Behavioural intention to decrease alcohol consumption will be measured with the question "I intend to cut down on the number of alcohol units that I drink in the forthcoming month" on 5-point Likert scale (Strongly Disagree to Strongly Agree), only at both follow-ups.
Emotional response to the labels | 1 week
  Emotional response to the labels will only be measured among those reporting to have noticed the labels: "Thinking about the labels on the alcohol containers I've seen as part of this study, I felt: disgusted / afraid / uncomfortable / worried" / excited / pleased" With Likert answers scale from 1 to 5 (1 = "not at all", 3 = "moderately", and 5 = "very").
Support for alcohol policies | 1 week / 1 month
  Support for alcohol policies will be measured with listing range of alcohol policies (e.g. increasing the price of alcohol, reducing the number of outlets that sell alcohol" and asking the participants "To what extent would you support the government in your country introducing the following alcohol-related policies? Please indicate your answer on the scale below from 1 (strongly disagree) to 5 (strongly agree).
Product appeal | 1 week
  It will only be measured among those reporting to have noticed the labels, with three items developed for this study ("I found the beverages less appealing after noticing the health information on the labels"; "The health information on the labels reduced my enjoyment of these beverages"; "I felt the health information on the label detracted from the overall alcohol product appearance") on 5-point Likert scale (Strongly Disagree to Strongly Agree).

CONTACTS AND LOCATIONS:
Overall Officials: Daša Kokole, PhD, Principal Investigator — World Health Organisation Regional Office for Europe
Locations (1):
- Sampled supermarkets in selected city neighbourhoods, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication(s).
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The dataset will be available following the open data sharing practices, and will be available on Figshare repository (https://figshare.com/) once the article with the main results is published.
Access Criteria: The interested researchers will be able to access and download the data directly through the platform, without requiring any permissions. The article, including the dataset will be shared under a noncommercial license (e.g. Creative Commons Attribution-NonCommercial (CC BY-NC)), allowing others to use the data for research, educational, or other noncommercial purposes, but not for commercial advantage or monetary gain.

REFERENCES:
- [Derived] Kokole D, Neufeld M, Correia D, Rehm J, Ferreira-Borges C, Hobin E, Rovira P, Segura Garcia L, Colom Farran J. Impacts of alcohol health warning labels in a real-world setting: protocol for a randomised controlled trial among supermarket customers in Barcelona. BMJ Open. 2026 Jan 21;16(1):e103464. doi: 10.1136/bmjopen-2025-103464. PMID 41565326